CLINICAL TRIAL: NCT01185002
Title: Evaluation of PillCam® Colon 2 Capsule Endoscopy Regimen
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MA-111
Record Dates: First submitted 2010-08-18; First posted 2010-08-19 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2011-02

CONDITIONS: Colonoscopy; Endoscopy
Keywords: CE; colonoscopy; colon; Eligable for colon evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- MgC boosts (Experimental): Subjects will be instructed to perform the colon preparation procedure and follow a detailed dietary regimen prior to and during the CE procedure.
  In this arm the subjects will be administered MgC boosts.
  Interventions: Other: PillCam® COLON 2 procedure using MgC boosts
- Suprep boosts (Experimental): Subjects will be instructed to perform the colon preparation procedure and follow a detailed dietary regimen prior to and during the CE procedure.
  In this arm the subjects will be administered Suprep boosts
  Interventions: Other: PillCam® COLON 2 procedure using Suprep boosts
- Suprep boosts - Reduced dose (Experimental): Subjects will be instructed to perform the colon preparation procedure and follow a detailed dietary regimen prior to and during the CE procedure.
  In this arm the subjects will be administered a reduced dose of Suprep boosts
  Interventions: Other: PillCam® COLON 2 procedure using reduced dose of Suprep boosts

INTERVENTIONS:
Other: PillCam® COLON 2 procedure using MgC boosts — Subjects will be instructed to perform the colon preparation procedure and follow a detailed dietary regimen prior to and during the CE procedure. During the CE procedure the subjects will be required to take MgC boosts.
  Arms: MgC boosts
Other: PillCam® COLON 2 procedure using Suprep boosts — Subjects will be instructed to perform the colon preparation procedure and follow a detailed dietary regimen prior to and during the CE procedure. During the CE procedure the subjects will be required to take Suprep boosts
  Arms: Suprep boosts
Other: PillCam® COLON 2 procedure using reduced dose of Suprep boosts — Subjects will be instructed to perform the colon preparation procedure and follow a detailed dietary regimen prior to and during the CE procedure. During the CE procedure the subjects will be required to take reduced dose of Suprep boosts
  Arms: Suprep boosts - Reduced dose

SUMMARY:
The purpose of the study is to test the effect of a bowel preparation and boosts regimen on PillCam® procedure, colon cleanliness and capsule excretion time.

DETAILED DESCRIPTION:
Interim analysis will be done after 20 subjects are enrolled in order to assess the 1st arm. Following the analysis of the first phase results, and per need, 30 more subjects may be enrolled under a different regimen (2nd arm). Second Interim analysis will be done in order to assess the 2nd phase results. Following the analysis of the 2nd phase results, and per need, up to 30 additional subjects may be enrolled under a third regimen (3rd arm).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 50 - 75 years of age.
2. Subject received an explanation about the nature of the study and agrees to provide written informed consent.

Exclusion Criteria:

1. Subject has dysphagia or any swallowing disorder
2. Subject has congestive heart failure
3. Subject has Diabetes type I.
4. Subject has had prior abdominal surgery other than uncomplicated procedures that would be unlikely to lead to bowel obstruction based on the clinical judgment of the investigator
5. Subject has a cardiac pacemaker or other implanted electro medical device.
6. Subject has any allergy or other known contraindication to the medications used in the study
7. Subject is expected to undergo MRI examination within 7 days after ingestion of the capsule.
8. Subject with any condition believed to have an increased risk for capsule retention such as Crohn's disease, intestinal tumors, radiation enteritis, and incomplete colonoscopies due to obstructions or NSAID enteropathy.
9. Subject with gastrointestinal motility disorders
10. Subject has known delayed gastric emptying
11. Subject has any condition, which precludes compliance with study and/or device instructions.
12. Women who are either pregnant or nursing at the time of screening, or are of child-bearing potential and do not practice medically acceptable methods of contraception.
13. Subject suffers from life threatening conditions
14. Subject currently participating in another clinical study

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Capsule excretion rate | 10 hours post capsule ingestion

SECONDARY OUTCOMES:
Distribution of PillCam® COLON 2 excretion times | Up to 12 hours and at least 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Rex, Prof., Principal Investigator — Division of Gastroenterology Indiana University Medical Center
Locations (7):
- United States (7):
  - Alabama Digestive Disorders Center, Huntsville, Alabama
  - Division of Gastroenterology Indiana University Medical Center, Indianapolis, Indiana
  - Research Associates of New York, New York, New York
  - University of North Carolina Division of Digestive Disease, Chapel Hill, North Carolina
  - Digestive Care, Inc., Beavercreek, Ohio
  - Franklin Gastroenterology, Franklin, Tennessee
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia